CLINICAL TRIAL: NCT01296750
Title: A Randomized Clinical Trial Comparing Late Versus Early Physiotherapy Start Times Following Multi Ligament Reconstruction for Knee Dislocation (Co-LEAP)
Brief Title: Late Compared to Early Physiotherapy Following Knee Dislocation
Acronym: Co_Leap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMH Co_LEAP
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2020-01

CONDITIONS: Traumatic Knee Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Physiotherapy (Active Comparator): Physiotherapy to begin within 1 day post op.
  Interventions: Other: Early Physiotherapy start
- Late Physiotherapy (No Intervention): Physiotherapy to start 6 weeks post op

INTERVENTIONS:
Other: Early Physiotherapy start — Physiotherapy starting at one day post op
  Arms: Early Physiotherapy

SUMMARY:
A knee dislocation is an unusual and extremely serious injury and is defined as complete displacement of the tibia with respect to the femur, usually with disruption of 3 or more of the stabilizing ligaments. When the knee dislocates, there is often significant damage to the soft-tissues envelope surrounding the joint, including adjacent neurovascular structures. Not surprisingly, this injury is a profoundly debilitating, life-altering event, with the potential to necessitate career change in athletes and laborers alike. Current evidence indicates that operative management for these injuries is more effective at returning patients to pre-morbid range of motion (ROM) and activity than conservative management. Post operative rehabilitation programs for these patients must balance the need for stability of their surgical repair and knee ROM and functionality. Experimental data suggests that post-operative immobilization offers greater protection of the surgical reconstruction, whereas immediate, aggressive physiotherapy may be more effective at preventing arthrofibrosis stiffness. The investigators are proposing a randomized clinical trial comparing early physiotherapy (day one post op) versus immobilization for three weeks then initiation of physiotherapy. The physiotherapy progams will be identicalbe in all aspects except for progam initiation.

ELIGIBILITY:
Inclusion Criteria:

* Ambulation without aids in pre-morbid condition
* Multi-ligament knee injury with or without associated peri-articular fracture
* Operative management within three weeks of the injury

Exclusion Criteria:

* Poly-trauma with life-threatening injuries preventing rehabilitation
* Patients unable to comply with intensive rehabilitation
* Patients unable or unlikely to maintain follow-up

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Need for knee manipulation at or within 6months of initial surgery. | 6 months
  Manipulation includes:
  1. Knee manipulation under anesthesia
  2. Arthroscopic debridement of arthrofibrosis
  3. Open debridement of arthrofibrosis

SECONDARY OUTCOMES:
Knee Range of Motion | 6 months
  Passive Range of Motion
Knee stability | 6 months
  Clinical exam of ligament grading
Patient Reported Outcome | 6 months
  Multi-Ligament Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hoit G, Rubacha M, Chahal J, Khan R, Ravi B, Whelan DB. Is There a Disadvantage to Early Physical Therapy After Multiligament Surgery for Knee Dislocation? A Pilot Randomized Clinical Trial. Clin Orthop Relat Res. 2021 Aug 1;479(8):1725-1736. doi: 10.1097/CORR.0000000000001729. PMID 33729214